CLINICAL TRIAL: NCT07204678
Title: Post Market Clinical Follow-up Study of the Precise Pro Rx Nitinol Stent System in the Treatment of Carotid Artery Disease (REAL-PRECISE)
Brief Title: PMCF Study of Precise Pro Rx for Carotid Artery Disease
Acronym: REAL-PRECISE
Status: Enrolling by invitation | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: Rede Optimus Hospitalar SA (Network)
Responsible Party: Sponsor
Other Study IDs: P21-7903
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid artery stenosis; PRECISE PRO Rx Nitinol Stent System
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects treated with the PRECISE PRO Rx Nitinol Stent System: Subjects treated with the PRECISE PRO Rx Nitinol Stent System according to the Instructions for Use for treatment of carotid artery stenosis
  Interventions: Device: PRECISE PRO Rx Nitinol Stent System

INTERVENTIONS:
Device: PRECISE PRO Rx Nitinol Stent System — The Cordis PRECISE PRO Rx Nitinol Stent System is a single-use device consisting of an endovascular stent and sheath delivery system, intended to deliver a self-expanding endovascular stent to the carotid artery(ies). The stent component imparts an outward radial force on the luminal surface of the vessel wall restoring vascular patency. The Cordis PRECISE PRO Rx Nitinol Stent System is indicated for use in patients with stenotic lesions of the carotid artery(ies).

SUMMARY:
The purpose of this study is to evaluate long-term clinical safety and performance of the PRECISE PRO RX Nitinol Stent System to treat stenotic lesions of the carotid arteries.

DETAILED DESCRIPTION:
The REAL-PRECISE study is a multi-center, non-randomized, observational analysis of retrospective data collected on subjects treated with PRECISE PRO Rx Nitinol Stent System. The purpose of this study is to evaluate the long-term (5-year) safety and performance of PRECISE PRO Rx Nitinol Stent System in subjects with stenotic lesions of the carotid arteries. The study is conducted in up to 15 European study sites in approximately 3 countries with high volume use of PRECISE PRO Rx. The enrollment and data collection takes approximately 4-6 months.

ELIGIBILITY:
NOTE: This is a RETROSPECTIVE study designed to collect outcomes on subjects who were already treated with the study device.

Inclusion Criteria:

* Subjects treated with the PRECISE PRO Rx Nitinol Stent System according to the Instructions for Use for treatment of carotid artery stenosis
* If an EC-approved informed consent waiver is not obtained, then documented informed consent from the subject or legal representative granting permission to share the subject's clinical data

Exclusion Criteria:

* Women who were pregnant or lactating at the time of the procedure
* Pediatric subjects (<18 years of age) at the time of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated with the PRECISE PRO Rx Nitinol Stent System according to the Instructions for Use for treatment of carotid artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Performance Endpoint - Technical Success | At the conclusion of the index procedure
  Achievement of a final residual stenosis of <30% at the target lesion using any percutaneous method at the conclusion of the index procedure
Performance Endpoint - Target Lesion Revascularization (TLR) at 12 months | At 12 months
  A repeat revascularization procedure performed at the original treatment site due to restenosis of ≥50% at the target lesion (as confirmed by quantitative angiography) in the presence of symptoms or ≥80% in the absence of symptoms
Safety Endpoint - All-Cause Mortality | Through 5 years
  All site-reported events of all-cause mortality
Safety Endpoint - Myocardial Infarction | Through 5 years.
  All site-reported events of myocardial infarction
Safety Endpoint - Major Stroke | Through 5 years
  A major stroke is defined as a cerebrovascular accident
Safety Endpoint - Minor Stroke | Through 5 years
  A minor stroke is defined as a transient ischemic attack
Safety Endpoint - Thrombosis | Through 5 years
  All site-reported events of thrombosis

OTHER OUTCOMES:
Stent Patency | Through 5 years
  The stent patency is defined as 30% stenosis immediately post-stent placement and < 50% stenosis long-term
All adverse events | Through 5 years
  All adverse events reported by sites
In-Stent Restenosis (ISR) | Through 5 years
  All site-reported events of In-Stent Restenosis (ISR) evaluated through any imaging assessment performed

CONTACTS AND LOCATIONS:
Overall Officials: Nusrath Sultana, Study Director — Cordis US Corp.
Locations (1):
- University Hospital Tulln, Tulln, Austria

IPD SHARING:
Plan to Share IPD: Undecided